CLINICAL TRIAL: NCT01265966
Title: Characterization of the Normal Cortisol Response to Moderate and Deep Sedation in Adrenally Sufficient Children
Brief Title: Cortisol Response to Moderate and Deep Sedation in Children
Status: Completed | Type: Observational
Sponsor: Tripler Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jordan Pinsker, Cheif, Pediatric Endocrinology, Tripler Army Medical Center
Other Study IDs: TAMC 32H10
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Adrenal Insufficiency
Keywords: Moderate Sedation; Sedation, Deep
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — This is an observational study measuring salivary cortisol levels. No interventions will done based on these measurements during the study. Specimens will be disposed off at the end of the study.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Moderate Sedation: Children undergoing moderate sedation for procedures.
- Deep Sedation: Children undergoing deep sedation for procedures.

SUMMARY:
Currently, it is unknown whether sedation itself induces a rise in serum cortisol levels or if cortisol levels rise under only the most invasive of procedures, regardless of the type of anesthetic agent used. Animal data shows significant alterations in steroid intermediates under anesthesia regardless of the procedure performed. Prior studies in children show general anesthesia and even epidural anesthesia can cause a rise in serum cortisol, but the effects of moderate and deep sedation on cortisol levels during different types of procedures are unknown. General medical practice varies considerably among providers; some provide stress dosing (extra and sometimes high doses of steroids) for sedation for both non-invasive and invasive procedures for patients with known adrenal insufficiency, but the doses given vary considerably. Others provide stress dosing only for the most invasive procedures in this population of patients. Currently there is no published normative data on changes in cortisol levels under moderate and deep sedation in adrenally sufficient children, so the normal response we are trying to mimic is unknown.

We propose to measure salivary cortisol levels prospectively in adrenally sufficient children undergoing moderate and deep sedation to determine the normal cortisol response to the stress of sedation for both invasive and non-invasive procedures.

Up to 300 adrenally sufficient children will be prospectively recruited to measure salivary cortisol levels during moderate and deep sedation for non-invasive procedures (e.g. MRI, echocardiogram, or other imaging studies), and invasive procedures (e.g. surgery, endoscopy) to determine what the normal cortisol response is to the stress of sedation during these procedures using various anesthetic agents.

The primary outcome variable will be to determine peak salivary cortisol measurements during non-invasive and invasive procedures under different levels of sedation using various anesthetic agents, and correlate these with known norms in children to determine if the patient's hypothalamic-pituitary-adrenal axis is under stress.

ELIGIBILITY:
Inclusion Criteria:

* Child presenting for routine sedation to the TAMC Pediatric Sedation Center.
* Age 3 months to 18 years of age.
* If female age 12 or greater OR menstruating, must not be pregnant.

Exclusion Criteria:

* Must not have the diagnosis of adrenal insufficiency or any concerns for possible adrenal insufficiency, to include recent tapering of exogenous steroids in the last 6 months.
* Current treatment with oral steroids or has been on oral steroids in the last 3 months.
* The use of regular inhaled corticosteroids for asthma controller treatment or intranasal steroids for allergic rhinitis is specifically NOT an exclusion criteria.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female military health care beneficiaries ages 3 months to 18 years of age presenting to the Tripler Army Medical Center pediatric sedation uni twho do not have any diagnosis consistent with or concerning for adrenal insufficiency, to include recent tapering of exogenous steroids in the last 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hsu, MD, Principal Investigator — Tripler Army Medical Center
Locations (1):
- Tripler Army Medical Center, Honolulu, Hawaii, United States

REFERENCES:
- [Result] Hsu AA, von Elten K, Chan D, Flynn T, Walker K, Barnhill J, Naun C, Pedersen AM, Ponaman M, Fredericks GJ, Crudo DF, Pinsker JE. Characterization of the cortisol stress response to sedation and anesthesia in children. J Clin Endocrinol Metab. 2012 Oct;97(10):E1830-5. doi: 10.1210/jc.2012-1499. Epub 2012 Aug 1. PMID 22855336

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited over a 7 month period from the Tripler Army Medical Center Pediatric Sedation Center.
Pre-assignment Details: 149 patients were recruited. 117 had samples adequate for analysis. 7 patients were on inhaled and/or intranasal steroids, and were analyzed separately. Therefore 110 were included in the main analysis.
Groups:
- General Anesthesia: Children undergoing general anesthesia for procedures.
Period: Overall Study
Arm/Group | Moderate Sedation | Deep Sedation | General Anesthesia
Started | 47 | 41 | 29
Analyzed Separately | 3 (Patients taking inhaled or intranasal corticosteroids were analyzed separately.) | 2 (Patients taking inhaled or intranasal corticosteroids were analyzed separately.) | 2 (Patients taking inhaled or intranasal corticosteroids were analyzed separately.)
Completed | 44 | 39 | 27
Not Completed | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Sedation | Deep Sedation | General Anesthesia | Total
Number analyzed (Participants) | 47 | 41 | 29 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 47 | 41 | 29 | 117
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 16 | 16 | 59
  Male | 20 | 25 | 13 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Peak Salivary Cortisol Level
Description: Salivary cortisol will be measured prior to the sedated procedure before any intravenous lines or other stress occurs, and then every 30 minutes into the sedated procedure while the patient is being routinely suctioned. Salivary cortisol will also be measured at the end of the procedure and 30 minutes post procedure (recovery). Because many different types of procedures are performed (imaging, endoscopy, surgical) the end times of the procedures will vary for each patient. The investigators will calculate a relative change from baseline for salivary cortisol levels by comparing the peak to baseline recorded level.
Time Frame: Baseline, then every 30 minutes, and at end of procedure
Population: All patients with adequate samples for analysis.
Measure: Mean (Standard Error); unit: Number (ratio of peak to baseline)
Arm/Group | Moderate Sedation | Deep Sedation | General Anesthesia
Number analyzed (Participants) | 44 | 39 | 27
Number (ratio of peak to baseline) | 2.9 (.2) | 4.3 (0.8) | 3.3 (1.0)

ADVERSE EVENTS:
Description: This was a minimal risk study. No adverse events for anticpated. No adverse events occured.
Arm/Group | Moderate Sedation | Deep Sedation | General Anesthesia
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/39 | 0/27
Other Adverse Events (participants affected / at risk) | 0/44 | 0/39 | 0/27

LIMITATIONS AND CAVEATS:
There is concern that the presence of a cortisol response is merely a biochemical phenomena and not of clinical importance for minor surgeries/mild stress.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No